CLINICAL TRIAL: NCT05533866
Title: Characterization of the Microbiome in Colonized Dystrophic and Junctional Epidermolysis Bullosa Wounds Before and After Use of APR-TD011 ® Spray Solution
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Amy Paller, Principal Investigator, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-5523
Record Dates: First submitted 2022-09-06; First posted 2022-09-09 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Epidermolysis Bullosa
MeSH Terms: conditions — Epidermolysis Bullosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- EB participants (Experimental): Visits will include screening, pre-treatment (week 0), weeks 4 and 8, followed by a visit without use of the APR-TD011 for 4 weeks (week 12) for microbiome assessment off of therapy.
  Interventions: Combination Product: APR-TD011

INTERVENTIONS:
Combination Product: APR-TD011 — APR-TD011 wound cleansing spray (drug/device combination product with a 510k clearance that is commercially marketed in the US for use by or on the order of a physician. Based on its product profile, APR-TD011 has been granted an FDA Orphan Drug Designation for epidermolysis bullosa.
  Other Names: Nexodyn AOS

SUMMARY:
In this pilot study, APR-TD011 antimicrobial wound cleansing spray will be given to all enrolled patients with junctional EB (JEB) or dystrophic epidermolysis bullosa (DEB) with Staphylococcus aureus or Pseudomonas aeruginosa culture-positive wounds. The primary aim will be to evaluate the change in skin microbiome (S. aureus, P. aeruginosa, commensal organisms) before, during, after treatment. Subjects who are colonized by S. aureus or pseudomonas will be treated for 8 weeks, will stop the spray and return at 12 weeks (4 weeks without the spray), and then will be able to use the spray as desired in a 6-month period of open-label use, with further feedback collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients 6 months of age or above with junctional or dystrophic epidermolysis bullosa
* Target wound that has been present for at least 3 weeks and is at least 10 cm2
* Target wound that is colonized with Staphylococcus aureus and/or Pseudomonas aeruginosa

Exclusion Criteria:

* Patients currently or recently (within past 4 weeks) on topical or systemic antibiotics
* Do not agree to avoid bathing or topical application at the target starting the night before the visit.
* Do not agree to avoid dilute bleach or vinegar baths, or other antiseptic use, at the target site starting at screening throughout the study.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2024-09-24 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Change in microbiome species | 8 weeks
  Reduction of Staphylococcus aureus between baseline and Week 8.

CONTACTS AND LOCATIONS:
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No